CLINICAL TRIAL: NCT02957682
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Praluent on Neurocognitive Function in Patients With Heterozygous Familial Hypercholesterolemia or With Non-Familial Hypercholesterolemia at High and Very High Cardiovascular Risk
Brief Title: Evaluating Effect of the Study Drug Praluent (Alirocumab) on Neurocognitive Function When Compared to Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R727-CL-1532; 2016-003189-16 (EudraCT Number)
Record Dates: First submitted 2016-10-28; First posted 2016-11-08 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Praluent Regimen - Administration through subcutaneous injection
  Interventions: Drug: Praluent (Alirocumab)
- Group 2 (Experimental): Placebo matching Praluent - Administration through subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Praluent (Alirocumab)
  Arms: Group 1
Drug: Placebo
  Arms: Group 2

SUMMARY:
The main purpose of this study is to evaluate the effect on mental state (known as "neurocognitive function") with use of Praluent.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women ≥ age 40 years and ≤ age 85 years
* Patients with heterozygous familial hypercholesterolemia (heFH) or with non-familial hypercholesterolemia (non-FH) patients at high or very high cardiovascular risk
* Patients with history of coronary heart disease (CHD) not having adequate control of their hypercholesterolemia with LDL-C ≥70 mg/dL, or all other patients with LDL-C ≥100 mg/dL and be on maximally-tolerated dose of statin (unless they are statin-intolerant)
* Patients must have successfully completed the Motor Screening Task
* Patients must be willing and able to comply with clinic visits and study related procedures
* Patients must provide signed informed consent

Key Exclusion Criteria:

* Patients with known Alzheimer's disease or other dementia, schizophrenia, bipolar disorder, severe depression, cognitive impairment, or patients with a sleep disorder requiring daily pharmacological treatment
* Recent (within 3 months prior to the screening visit) myocardial infarction, unstable angina leading to hospitalization, coronary artery bypass graft surgery, percutaneous coronary intervention, uncontrolled cardiac arrhythmia, carotid surgery or stenting, stroke, transient ischemic attack, carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease
* Certain laboratory findings obtained during the screening visit as defined in the protocol
* Any condition or situation, including other significant mental or neurological disorders that, in the investigator's opinion, may confound the study results, or may interfere significantly with the patient's participation in the study
* Pregnant or breastfeeding women
* A positive human immunodeficiency virus (HIV) test

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2176 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (147):
- United States (67):
  - Regeneron Study Site, Auburn, Alabama
  - Regeneron Study Site, Birmingham, Alabama
  - Regeneron Study Site, Mobile, Alabama
  - Regeneron Study Site, Beverly Hills, California
  - Regeneron Study Site, Los Gatos, California
  - Regeneron Study Site, North Hollywood, California
  - Regeneron Study Site, Port Hueneme, California
  - Regeneron Study Site, Westminster, California
  - Regeneron Study Site 1, Aurora, Colorado
  - Regeneron Study Site 2, Aurora, Colorado
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Lake Worth, Florida
  - Regeneron Study Site, Miami Springs, Florida
  - Regeneron Study Site, Covington, Georgia
  - Regeneron Study Site, Champaign, Illinois
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Rock Island, Illinois
  - Regeneron Study Site, Evansville, Indiana
  - Regeneron Study Site, Indianapolis, Indiana
  - Regeneron Study Site, Ames, Iowa
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, Waterloo, Iowa
  - Regeneron Study Site, Hutchinson, Kansas
  - Regeneron Study Site, Newton, Kansas
  - Regeneron Study Site, Overland Park, Kansas
  - Regeneron Study Site, Louisville, Kentucky
  - Regeneron Study Site, Bangor, Maine
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Oxon Hill, Maryland
  - Regeneron Study Site, Minneapolis, Minnesota
  - Regeneron Study Site, Olive Branch, Mississippi
  - Regeneron Study Site, Washington, Missouri
  - Regeneron Study Site, Buffalo, New York
  - Regeneron Study Site, New Hyde Park, New York
  - Regeneron Study Site, Cary, North Carolina
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Greensboro, North Carolina
  - Regeneron Study Site, Hickory, North Carolina
  - Regeneron Study Site, High Point, North Carolina
  - Regeneron Study Site, Raleigh, North Carolina
  - Regeneron Study Site, Rocky Mount, North Carolina
  - Regeneron Study Site, Salisbury, North Carolina
  - Regeneron Study Site, Statesville, North Carolina
  - Regeneron Study Site, Wilmington, North Carolina
  - Regeneron Study Site, Winston-Salem, North Carolina
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Cleveland, Ohio
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Duncansville, Pennsylvania
  - Regeneron Study Site, Charleston, South Carolina
  - Regeneron Study Site, Greenville, South Carolina
  - Regeneron Study Site, Summerville, South Carolina
  - Regeneron Study Site, Rapid City, South Dakota
  - Regeneron Study Site, Bristol, Tennessee
  - Regeneron Study Site, Knoxville, Tennessee
  - Regeneron Study Site, Powell, Tennessee
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Schertz, Texas
  - Regeneron Study Site, Shavano Park, Texas
  - Regeneron Study Site, Falls Church, Virginia
  - Regeneron Study Site, Winchester, Virginia
  - Regeneron Study Site, Burien, Washington
  - Regeneron Study Site, Everett, Washington
  - Regeneron Study Site, Tacoma, Washington
  - Regeneron Study Site, Walla Walla, Washington
  - Regeneron Study Site, Manitowoc, Wisconsin
- Bulgaria (6):
  - Regeneron Study Site, Pleven
  - Regeneron Study Site, Plovdiv
  - Regeneron Study Site, Sofia
  - Regeneron Study Site, Stara Zagora
  - Regeneron Study Site 1, Varna
  - Regeneron Study Site 2, Varna
- Chile (5):
  - Regeneron Study Site, Osorno
  - Regeneron Study Site, San Miguel
  - Regeneron Study Site, Santiago
  - Regeneron Study Site, Temuco
  - Regeneron Study Site, Viña del Mar
- Estonia (5):
  - Regeneron Study Site, Paide
  - Regeneron Study Site, Tallinn
  - Regeneron Study Site 1, Tallinn
  - Regeneron Study Site 2, Tallinn
  - Regeneron Study Site, Tartu
- Japan (12):
  - Regeneron Study Site, Nishinomiya, Hogo
  - Regeneron Study Site, Kahoku-gun, Ishikawa-ken
  - Regeneron Study Site, Kawasaki, Kanagawa
  - Regeneron Study Site, Yokohama, Kanagawa
  - Regeneron Study Site, Uji-shi, Kyoto
  - Regeneron Study Site, Nakagami-gun, Okinawa
  - Regeneron Study Site, Iruma-gun, Saitama
  - Regeneron Study Site, Bunkyō-Ku, Tokyo
  - Regeneron Study Site, Chuo Ku, Tokyo
  - Regeneron Study Site, Hachiōji, Tokyo
  - Regeneron Study Site, Itabashi-ku, Tokyo
  - Regeneron Study Site, Shinagawa-Ku, Tokyo
- Mexico (15):
  - Regeneron Study Site, Aguascalientes
  - Regeneron Study Site, Cuernavaca
  - Regeneron Study Site, Culiacán
  - Regeneron Study Site, Distrito Federal
  - Regeneron Study Site, Durango
  - Regeneron Study Site, Guadalajara
  - Regeneron Study Site, Mexico City
  - Regeneron Study Site, Mérida
  - Regeneron Study Site 1, Monterrey
  - Regeneron Study Site 2, Monterrey
  - Regeneron Study Site, Monterrey
  - Regeneron Study Site, Pachuca
  - Regeneron Study Site, Querétaro
  - Regeneron Study Site, San Juan del Río
  - Regeneron Study Site, Torreón
- Russia (11):
  - Regeneron Study Site, Ivanovo
  - Regeneron Study Site, Kirov
  - Regeneron Study Site, Moscow
  - Regeneron Study Site, Novosibirsk
  - Regeneron Study Site, Rostov-on-Don
  - Regeneron Study Site, Saint Petersburg
  - Regeneron Study Site, Saratov
  - Regeneron Study Site, Tyumen
  - Regeneron Study Site, Yaroslavl
  - Regeneron Study Site 1, Yaroslavl
  - Regeneron Study Site 2, Yaroslavl
- South Africa (15):
  - Regeneron Study Site, Kuils River, Cape Town
  - Regeneron Study Site, Port Elizabeth, Eastern Cape
  - Regeneron Study Site, Halfway House, Gauteng
  - Regeneron Study Site, Pretoria, Gauteng
  - Regeneron Study Site, Pretoria West, Gauteng
  - Regeneron Study Site, Kempton Park, Johannesburg
  - Regeneron Study Site, Soweto, Johannesburg
  - Regeneron Study Site, Middelburg, Mpumalanga
  - Regeneron Study Site, Cape Town, Western Cape
  - Regeneron Study Site, Paarl, Western Cape
  - Regeneron Study Site, Somerset West, Western Cape
  - Regeneron Study Site, Worcester, Western Cape
  - Regeneron Study Site 1, Bloemfontein
  - Regeneron Study Site 2, Bloemfontein
  - Regeneron Study Site, Claremont
- Ukraine (11):
  - Regeneron Study Site, Uzhhorod, Transcarpathian Region
  - Regeneron Study Site, Kharkiv
  - Regeneron Study Site 1, Kiev
  - Regeneron Study Site 2, Kiev
  - Regeneron Study Site, Kyiv
  - Regeneron Study Site 1, Kyiv
  - Regeneron Study Site 2, Kyiv
  - Regeneron Study Site, Lviv
  - Regeneron Study Site 1, Vinnitsa
  - Regeneron Study Site 2, Vinnitsa
  - Regeneron Study Site, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2176 participants were randomized across 169 sites in Bulgaria, Chile, Estonia, Japan, Mexico, Russian Federation, South Africa, Ukraine, and the United States
Pre-assignment Details: Participants who met the eligibility criteria were randomized in 1:1 ratio into 2 treatment groups: placebo and alirocumab. Randomization was stratified by age (less than [<] 65 or greater than or equal to [>=] 65) and by statin use (no statin, low lipophilicity of the concomitant statin, or high lipophilicity of the concomitant statin).
Groups:
- Placebo: Participants received subcutaneous (SC) injections of placebo matched to alirocumab every 2 weeks (Q2W) up to 94 weeks.
- Alirocumab 75 Q2W/Up150 Q2W: Participants received SC injections of alirocumab at a dose of 75 milligrams (mg) Q2W and up-titrated to 150 mg Q2W at Week 12 in a blinded fashion (if LDL-C ≥ 50 mg/dL at Week 8) up to 94 weeks.
Period: Overall Study
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Started (Randomized) | 1088 | 1088
Randomized and Treated | 1085 | 1086
Completed (Completed 96-week study treatment period) | 890 | 919
Not Completed | 198 | 169
Not completed — Adverse Event | 64 | 67
Not completed — Poor Compliance to Protocol | 30 | 26
Not completed — Physician Decision | 4 | 4
Not completed — Study Terminated by Sponsor | 4 | 3
Not completed — Subject Moved | 10 | 16
Not completed — Withdrawal by Subject | 64 | 33
Not completed — Related to IMP Administration | 3 | 6
Not completed — Non-disclosed | 16 | 12
Not completed — Discontinued After Randomization and Prior to Any Treatment | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety population (SAF) included all participants randomized and exposed to at least one dose of study drug, regardless of the amount of treatment administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W | Total
Number analyzed (Participants) | 1084 | 1087 | 2171
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (9.02) | 62.6 (8.88) | 62.6 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 459 | 448 | 907
  Male | 625 | 639 | 1264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 137 | 142 | 279
  Not Hispanic or Latino | 945 | 943 | 1888
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 888 | 886 | 1774
    Black or African American | 86 | 77 | 163
    Asian | 19 | 28 | 47
    American Indian or Alaska Native | 11 | 16 | 27
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Other | 80 | 80 | 160
CANTAB Cognitive Domain Spatial Working Memory (SWM) Strategy Raw Score [Mean (Standard Deviation); unit: Units on a Scale] — Cambridge Neuropsychological Test Automated Battery (CANTAB) SWM task assessed cognitive domain of executive function. Colored boxes were shown on a screen. A token was hidden in one of the boxes (never same box twice). Instructions were to touch boxes to search for token until number of tokens found equaled number of boxes. SWM strategy index represents number of times a search began with a different box. Baseline SWM strategy score is the last score obtained before first dose of study treatment. Raw score ranges from 4 to 28. A high score represents inefficient use of strategy. Population: Primary safety population included participants from the safety population who had an assessment of the SWM strategy score at baseline (the last score obtained before the first dose of study treatment) and at least 1 score measured during the Treatment-Emergent Adverse Event (TEAE) period.
  Units on a Scale
    number analyzed (Participants) | 1035 | 1051 | 2086
    (all) | 15.9 (5.03) | 16.05 (5.11) | 16.0 (5.07)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cambridge Neuropsychological Test Automated Battery (CANTAB) Cognitive Domain Spatial Working Memory (SWM) Strategy Z-Score at Week 96
Description: CANTAB SWM task assessed cognitive domain of executive function. Colored boxes were shown on a screen. A token was hidden in one of the boxes (never same box twice). Instructions were to touch boxes to search for token until number of tokens found equaled number of boxes. SWM strategy index represents number of times a search began with a different box. Z-score represents standardized measure of how far an individual deviated from study cohort average at baseline. A higher Z-score reflects better performance.
Time Frame: Week 96
Population: Primary safety population included participants from the safety population who had an assessment of the SWM strategy score at baseline, and at least 1 score measured during the treatment-emergent adverse event (TEAE) period. The TEAE period is defined as the first double-blind treatment dose to last dose of double-blind treatment + 70 days (10 weeks). Participants were analyzed according to the treatment actually received.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1035 | 1051
Z-score | -0.180 (0.027) | -0.200 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 Q2W/Up150 Q2W; Change at Week 96; Test type: Non-Inferiority — Upper confidence interval (CI) limit was compared to the noninferiority margin, which was 0.2%, and noninferiority was declared if the upper CI limit was below the noninferiority margin; p = 0.6055, Mixed-effect Model Repeated Measures — P-value was taken from mixed-effect model with repeated measures (MMRM) analysis; Least Square (LS) Mean Difference = -0.020, 95% CI 2-sided [-0.094 to 0.055] — Model: fixed categorical effects of treatment group, randomization strata as per IVRS, time point, treatment-by-time point, strata-by-time point, continuous fixed covariates of baseline SWMS raw score value, baseline value by time-point interaction

2. Secondary Outcome: Change From Baseline in CANTAB Cognitive Domain SWM Strategy Raw Score at Week 96
Description: CANTAB SWM task assessed cognitive domain of executive function. Colored boxes were shown on a screen. A token was hidden in one of the boxes (never same box twice). Instructions were to touch boxes to search for token until number of tokens found equaled number of boxes. SWM strategy index represents number of times a search began with a different box. Lower change from baseline raw scores reflect better SWM performance (i.e. less impairment).
Time Frame: Week 96
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1035 | 1051
Units on a Scale | -0.9 (4.49) | -1.0 (4.31)

3. Secondary Outcome: Percent Change From Baseline in Calculated Low-density Lipoprotein Cholesterol (LDL-C) at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in calculated LDL-C at Week 12, 24, 48, 72, and 96 was reported. LDL-C was measured using conventional units milligram per deciliter (mg/dL).
Time Frame: Week 12, 24, 48, 72, and 96
Population: Intent-to-treat (ITT) population included all participants with availability of at least 1 measurement value for calculated LDL-C before first dose of study drug (i.e. baseline) and within 1 of the analysis windows during the main efficacy period; the main efficacy period is defined as the time from the first double-blind study treatment injection up to the upper limit of the week 96 analysis window. ITT population analyzed according to treatment group allocated by randomization (as-randomized).
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | 0.6 (1.0) | -49.6 (0.9)
  Percent change at Week 24 | 3.0 (1.0) | -54.2 (1.0)
  Percent change at Week 48 | 2.8 (1.1) | -51.4 (1.1)
  Percent change at Week 72 | 2.4 (1.2) | -50.4 (1.2)
  Percent change at Week 96 | 4.0 (1.3) | -46.2 (1.3)

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in Apo B at Week 12, 24, 48, 72, and 96 was reported. Apo B was measured using conventional units mg/dL.
Time Frame: Week 12, 24, 48, 72, and 96
Population: ITT population included all participants with availability of at least 1 measurement value for calculated LDL-C before first dose of study drug (i.e. baseline) and within 1 of the analysis windows during the main efficacy period; the main efficacy period is defined as the time from the first double-blind study treatment injection up to the upper limit of the week 96 analysis window. ITT population analyzed according to treatment group allocated by randomization (as-randomized).
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | 0.8 (0.7) | -36.7 (0.7)
  Percent change at Week 24 | 2.1 (0.8) | -40.9 (0.8)
  Percent change at Week 48 | 1.1 (0.8) | -39.0 (0.8)
  Percent change at Week 72 | 0.2 (0.9) | -39.1 (0.8)
  Percent change at Week 96 | 1.4 (0.9) | -36.4 (0.9)

5. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in non-HDL-C at Week 12, 24, 48, 72, and 96 was reported. Non-HDL-C was measured using conventional units mg/dL.
Time Frame: Week 12, 24, 48, 72, and 96
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | 0.7 (0.8) | -40.4 (0.8)
  Percent change at Week 24 | 2.2 (0.9) | -44.0 (0.9)
  Percent change at Week 48 | 1.7 (0.9) | -41.1 (0.9)
  Percent change at Week 72 | 1.7 (1.0) | -40.6 (1.0)
  Percent change at Week 96 | 2.5 (1.1) | -37.0 (1.1)

6. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in calculated Total-C at Week 12, 24, 48, 72, and 96 was reported. Total-C was measured using conventional units mg/dL.
Time Frame: Week 12, 24, 48, 72, and 96
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | -0.3 (0.6) | -29.6 (0.6)
  Percent change at Week 24 | 1.5 (0.6) | -31.8 (0.6)
  Percent change at Week 48 | 1.1 (0.7) | -29.6 (0.7)
  Percent change at Week 72 | 1.1 (0.7) | -29.0 (0.7)
  Percent change at Week 96 | 1.8 (0.7) | -26.5 (0.7)

7. Secondary Outcome: Percent Change From Baseline in Lipoprotein a [Lp(a)] at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in Lp(a) at Week 12, 24, 48, 72, and 96 was reported. Lp(a) was measured using conventional units mg/dL.
Time Frame: Week 12, 24, 48, 72, and 96
Population: ITT Population was used. The two-step multiple imputation procedure is used to address missing values in the randomized population. In the first step, the monotone missing pattern is induced in the multiply-imputed data. In the second step, the missing data at subsequent visits are imputed using the regression method for continuous variables.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | -3.3 (0.8) | -22.4 (0.8)
  Percent change at Week 24 | -0.5 (0.9) | -24.7 (0.9)
  Percent change at Week 48 | -1.4 (1.0) | -24.3 (1.0)
  Percent change at Week 72 | -1.7 (1.0) | -25.1 (1.0)
  Percent change at Week 96 | 4.8 (1.1) | -17.7 (1.1)

8. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in HDL-C at Week 12, 24, 48, 72, and 96 was reported. HDL-C was measured using conventional units mg/dL.
Time Frame: Week 12, 24, 48, 72, and 96
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | 0.6 (0.5) | 5.9 (0.5)
  Percent change at Week 24 | 3.8 (0.6) | 9.0 (0.6)
  Percent change at Week 48 | 3.8 (0.6) | 9.2 (0.6)
  Percent change at Week 72 | 4.4 (0.7) | 10.3 (0.6)
  Percent change at Week 96 | 5.5 (0.7) | 10.8 (0.7)

9. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in TG at Week 12, 24, 48, 72, and 96 was reported. TG was measured using conventional units mg/dL.
Time Frame: Week 12, 24, 48, 72, and 96
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | 0.7 (1.0) | -11.0 (1.0)
  Percent change at Week 24 | -1.8 (1.0) | -12.9 (1.0)
  Percent change at Week 48 | -1.8 (1.1) | -11.3 (1.1)
  Percent change at Week 72 | -2.1 (1.1) | -12.3 (1.1)
  Percent change at Week 96 | -2.7 (1.1) | -11.9 (1.1)

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) A-1 at Week 12, 24, 48, 72, and 96
Description: Percent change from baseline in Apo A-1 at Week 12, 24, 48, 72, and 96 was reported. Apo A-1 was measured using conventional units mg/dL.
Time Frame: Week 12, 24, 48, 72, and 96
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percent Change
  Percent change at Week 12 | -1.3 (0.4) | 1.7 (0.4)
  Percent change at Week 24 | 2.9 (0.4) | 6.1 (0.4)
  Percent change at Week 48 | 4.7 (0.4) | 7.7 (0.4)
  Percent change at Week 72 | 4.4 (0.4) | 7.8 (0.4)
  Percent change at Week 96 | 4.2 (0.4) | 7.5 (0.4)

11. Secondary Outcome: Percentage of Participants Who Reached Low Density Lipoprotein Cholesterol (LDL-C) Level Less Than (<) 70 mg/dL (1.81 Millimoles Per Liter [mmol/L]) at Week 12, 24, 48, 72, and 96
Description: Percentage of participants who reached LDL-C level < 70 mg/dL (1.81 mmol/L) at Week 12, 24, 48, 72, and 96 were reported.
Time Frame: Week 12, 24, 48, 72, and 96
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percentage of Participants
  Week 12 | 10.3 | 69.4
  Week 24 | 8.4 | 74.7
  Week 48 | 10.7 | 71.4
  Week 72 | 11.3 | 69.7
  Week 96 | 10.7 | 64.5

12. Secondary Outcome: Percentage of Participants Who Reached Low Density Lipoprotein Cholesterol (LDL-C) Level Less Than (<) 50 mg/dL (1.29 mmol/L) at Week 12, 24, 48, 72, and 96
Description: Percentage of participants who reached LDL-C level < 50 mg/dL (1.29 mmol/L) at Week 12, 24, 48, 72, and 96 were reported.
Time Frame: Week 12, 24, 48, 72, and 96
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1051 | 1058
Percentage of Participants
  Week 12 | 1.7 | 45.6
  Week 24 | 2.0 | 56.9
  Week 48 | 2.1 | 51.3
  Week 72 | 2.5 | 52.1
  Week 96 | 2.4 | 46.4

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. TEAE was defined as AEs that developed or worsened/became serious during on-treatment period (time from the first double-blind study treatment injection up to 70 days after the last double-blind study treatment injection). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-participant hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Up to Week 96
Population: Safety population included all participants randomized and exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1084 | 1087
Participants
  Participants with any TEAEs | 857 | 866
  Participants with any Serious TEAEs | 216 | 189
  Participants with any TEAE leading to death | 17 | 13
  Participants with any TEAE leading to permanent treatment discontinuation | 59 | 64

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the end of study (Week 96) regardless of seriousness or relationship to investigational product (IP).
Description: Safety population included all participants randomized and exposed to at least one dose of study drug, regardless of the amount of treatment administered. Participants were analyzed according to the treatment received (placebo or Praluent 75 mg Q2W/up-titrate 150 mg Q2W).
Arm/Group | Placebo | Alirocumab 75 Q2W/Up150 Q2W
All-Cause Mortality (participants affected / at risk) | 24/1084 | 17/1087
Serious Adverse Events (participants affected / at risk) | 216/1084 | 189/1087
Other Adverse Events (participants affected / at risk) | 387/1084 | 366/1087
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1084) | Alirocumab 75 Q2W/Up150 Q2W (N=1087)
Angina unstable (Cardiac disorders) | 16 (17) | 14 (17)
Atrial fibrillation (Cardiac disorders) | 13 (16) | 5 (5)
Angina pectoris (Cardiac disorders) | 10 (12) | 11 (11)
Coronary artery disease (Cardiac disorders) | 8 (8) | 6 (8)
Acute myocardial infarction (Cardiac disorders) | 7 (7) | 5 (5)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4) | 4 (4)
Myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 4 (4)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (4)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Frederick's syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (8) | 6 (6)
Aortic aneurysm (Vascular disorders) | 3 (3) | 1 (1)
Hypertensive crisis (Vascular disorders) | 3 (4) | 3 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 2 (2)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Paget-Schroetter syndrome (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3) | 4 (4)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue haemorrhagic fever (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Haemorrhagic fever with renal syndrome (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acinic cell carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of epididymis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 5 (5) | 4 (4)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 3 (3)
Sciatica (Nervous system disorders) | 2 (3) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Multifocal motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oroantral fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Strangulated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2)
Chest pain (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Medical device site haematoma (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 2 (2)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 4 (4)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vestibulocerebellar syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Homicide (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1084) | Alirocumab 75 Q2W/Up150 Q2W (N=1087)
Bronchitis (Infections and infestations) | 65 (72) | 60 (78)
Influenza (Infections and infestations) | 69 (77) | 63 (69)
Nasopharyngitis (Infections and infestations) | 89 (117) | 82 (98)
Urinary tract infection (Infections and infestations) | 46 (65) | 61 (78)
Back pain (Musculoskeletal and connective tissue disorders) | 71 (82) | 60 (66)
Headache (Nervous system disorders) | 85 (123) | 71 (83)
Hypertension (Vascular disorders) | 73 (93) | 64 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02957682/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02957682/SAP_001.pdf